CLINICAL TRIAL: NCT03538535
Title: Computational Modeling of Reinforcement Learning in Depression
Brief Title: Set Your Goal: Engaging Go/No-Go Active Learning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00206862
Record Dates: First submitted 2018-05-14; First posted 2018-05-29 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Depression; Anxiety
Keywords: reinforcement learning; computational models; neuroimaging
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Adapted version of Behavioral Activation psychotherapy designed to optimize decision making and learning.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Go/No-Go Active Learning (GOAL) (Experimental): Adaptation of Behavioral Activation, focused on reinforcement learning strategies.
  Interventions: Behavioral: Go/No-Go Active Learning (GOAL)

INTERVENTIONS:
Behavioral: Go/No-Go Active Learning (GOAL) — Behavioral Activation psychotherapy adapted to engage go/no-go learning

SUMMARY:
This study will test a computational model reinforcement learning in depression and anxiety and test the extent to which the computational model predicts response to an adapted version of behavioral activation psychotherapy. The model will be based on a data from a computer task of reinforcement learning during 3T functional magnetic resonance imaging at baseline.

DETAILED DESCRIPTION:
The dysfunction of reinforcement learning is emerging as a transdiagnostic dimension of mood and anxiety. Computational models of reinforcement learning may expedite our ability to identify predictors of response, thereby improving efficacy rates. We will will, first, examine the neural substrates of reinforcement learning in depression and anxiety, and, second, test a computational model of reinforcement learning as a predictor of response to an adapted version of behavioral activation psychotherapy. Subjects (N=10) will be enrolled in a two week evaluation, followed with a nine week weekly intervention program. Assessments will be conducted at baseline, and during the intervention as the 3-, 6-, 9-week follow-ups. Reinforcement learning will be measured using 3T magnetic resonance imaging during a computer task. All other measures include structured clinical interviews, questionnaires, and computer tasks.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 21 and 40
* Physically healthy
* Right handed
* Normal or corrected to normal vision
* Scores equal or higher of (a) 24 on Inventory of Depressive Symptomatology, Self Report, or (b) 15 on the Generalized Anxiety Disorder Self Report.

Exclusion Criteria:

* Not currently in therapy or taking medications for anxiety or depression
* No contraindications for the magnetic resonance scan (claustrophobic)
* No history of head trauma, seizures, loss of consciousness
* Not taking hormone replacement, not pregnant
* No imminent suicidality
* No report of excessive alcohol or drug use in past three months

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Integrated Bayesian Information Criterion (BIC) score based on models using modified Q-learning models with two pairs of action values (go and no-go) for each state. | Baseline (Week 0)
  Models will include a learning rate, a slope of the softmax rule, noise factor, a bias factor to the action-value for 'go', and a Pavlovian factor.

CONTACTS AND LOCATIONS:
Overall Officials: Jackie Gollan, Ph.D., Principal Investigator — Associate Professor of Psychiatry and Behavioral Science
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huys QJM, Russek EM, Abitante G, Kahnt T, Gollan JK. Components of Behavioral Activation Therapy for Depression Engage Specific Reinforcement Learning Mechanisms in a Pilot Study. Comput Psychiatr. 2022 Oct 13;6(1):238-255. doi: 10.5334/cpsy.81. eCollection 2022. PMID 38774780